CLINICAL TRIAL: NCT00369486
Title: A Pilot Study of Peribulbar Triamcinolone Acetonide for Diabetic Macular Edema
Acronym: Peribulbar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Director, Jaeb Center for Health Research (DRCR.net)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEI-104; U10EY018817-03 (NIH); U10EY014229-07 (NIH); U10EY014231-09 (NIH)
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic; macular; edema; peribulbar; triamcinolone; acetonide; laser; photocoagulation; intraocular; DME
MeSH Terms: conditions — Edema | interventions — Triamcinolone; Triamcinolone Acetonide; Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): Focal laser photocoagulation (modified Early Treatment Diabetic Retinopathy Study (ETDRS) technique)
  Interventions: Procedure: Focal laser photocoagulation
- 2 (Experimental): Posterior peribulbar injection of 40 mg triamcinolone (Kenalog)
  Interventions: Drug: 40mg triamcinolone
- 3 (Experimental): Anterior peribulbar injection of 20 mg triamcinolone
  Interventions: Drug: 20mg triamcinolone
- 4 (Experimental): Posterior peribulbar injection of 40 mg triamcinolone followed after one month by laser
  Interventions: Drug: 40mg triamcinolone + laser
- 5 (Experimental): Anterior peribulbar injection of 20 mg triamcinolone followed after one month by laser
  Interventions: Drug: 20mg triamcinolone + laser

INTERVENTIONS:
Procedure: Focal laser photocoagulation — Focal laser photocoagulation (modified Early Treatment Diabetic Retinopathy Study technique)
  Other Names: focal/grid laser
  Arms: 1
Drug: 40mg triamcinolone — Posterior peribulbar injection of 40 mg triamcinolone (Kenalog)
  Other Names: Kenalog
  Arms: 2
Drug: 20mg triamcinolone — Anterior peribulbar injection of 20 mg triamcinolone
  Other Names: Kenalog
  Arms: 3
Drug: 40mg triamcinolone + laser — Posterior peribulbar injection of 40 mg triamcinolone followed after one month by laser
  Other Names: Kenalog; focal/grid photocoagulation
  Arms: 4
Drug: 20mg triamcinolone + laser — Anterior peribulbar injection of 20 mg triamcinolone followed after one month by laser
  Other Names: Kenalog; focal/grid photocoagulation
  Arms: 5

SUMMARY:
The study involves the enrollment of patients over 18 years of age with diabetic macular edema involving the center of the macula who have not already been given maximal laser treatment.

Patients with one study eye will be randomly assigned (stratified by prior laser) with equal probability to one of five treatment groups:

1. Focal laser photocoagulation (modified ETDRS technique)
2. Posterior peribulbar injection of 40 mg triamcinolone (Kenalog)
3. Anterior peribulbar injection of 20 mg triamcinolone
4. Posterior peribulbar injection of 40 mg triamcinolone followed after one month by laser
5. Anterior peribulbar injection of 20 mg triamcinolone followed after one month by laser

For patients with two study eyes (both eyes eligible at the time of randomization), the right eye (stratified by prior laser) will be randomly assigned with equal probabilities to one of the five treatment groups listed above. If the right eye was assigned to laser only, then the left eye will be assigned to one of the four triamcinolone groups above with equal probability (stratified by prior laser). If the right eye was assigned to receive triamcinolone, then the left eye will receive laser only.

Triamcinolone acetonide will be the corticosteroid utilized in this study. The triamcinolone acetonide preparation to be used is Kenalog. Kenalog is manufactured by Bristol Myers Squibb and is approved by the Food and Drug Administration for intramuscular use for a variety of indications. Peribulbar injections of Kenalog have been used for a wide variety of ocular conditions, particularly uveitis and post-cataract extraction cystoid macular edema, for many years.

Two different triamcinolone regimens will be assessed in the study: 40 mg injected posteriorly and 20 mg injected anteriorly. There is no indication of which treatment regimen will be better. Although the injection behind the eye is more common than the injection near the front of the eye, the injection near the front of the eye has less risk of injuring the eye. However, it is possible that the injection near the front of the eye may increase eye pressure more frequently. Little is known about which of the two injections decreases macular edema and improves vision more often.

Patients enrolled into the study will be followed for three years and will have study visits 1 month, 2 months, 4 months, 8 months and annually after receiving their assigned study treatment. For the first 8 months of the study, patients should only be retreated with their randomized treatment. However, if the patient's visual acuity has decreased by 15 letters or more, then any treatment may be given at the investigator's discretion. After completion of the 8-month visit, treatment is at investigator discretion.

The primary objective of this study is to obtain estimates of efficacy and safety outcomes for each of the treatment groups. These estimates will provide a basis for the sample size estimation and hypothesis generation in a phase III trial.

DETAILED DESCRIPTION:
Diabetic retinopathy is a major cause of visual impairment in the United States. Diabetic macular edema (DME) is a manifestation of diabetic retinopathy that produces loss of central vision. Data from the Wisconsin Epidemiologic Study of Diabetic Retinopathy (WESDR) estimate that after 15 years of known diabetes, the prevalence of diabetic macular edema is approximately 20% in patients with type 1 diabetes mellitus (DM), 25% in patients with type 2 DM who are taking insulin, and 14% in patients with type 2 DM who do not take insulin.

Diabetic macular edema results from abnormal leakage of macromolecules, such as lipoproteins, from retinal capillaries into the extravascular space followed by an oncotic influx of water into the extravascular space. Abnormalities in the retinal pigment epithelium may also cause or contribute to diabetic macular edema. These abnormalities may allow increased fluid from the choriocapillaries to enter the retina or they may decrease the normal efflux of fluid from the retina to the choriocapillaris. The mechanism of breakdown of the blood retina barrier at the level of the retinal capillaries and the retinal pigment epithelium may be due to changes to tight junction proteins such as occludin.

The increase in retinal capillary permeability and subsequent retinal edema may be the result of a breakdown of the blood retina barrier mediated in part by vascular endothelial growth factor (VEGF), a 45 kD glycoprotein. Aiello et al, demonstrated in an in vivo model that VEGF can increase vascular permeability. Fifteen eyes of 15 albino Sprague-Dawley rats received an intravitreal injection of VEGF. The effect of intravitreal administration of VEGF on retinal vascular permeability was assessed by vitreous fluorophotometry. In all 15 eyes receiving an intravitreal injection of VEGF, a statistically significant increase in vitreous fluorescein leakage was recorded. In contrast, control eyes, which were fellow eyes injected with vehicle alone, did not demonstrate a statistically significant increase in vitreous fluorescein leakage. Vitreous fluorescein leakage in eyes injected with VEGF attained a maximum of 227% of control levels.

Antonetti et al, demonstrated that VEGF may regulate vessel permeability by increasing phosphorylation of tight junction proteins such as occludin and zonula occluden 1. Sprague-Dawley rats were given intravitreal injections of VEGF and changes in tight junction proteins were observed through Western blot analysis. Treatment with alkaline phosphatase revealed that these changes were caused by a change in phosphorylation of tight junction proteins. This model provides, at the molecular level, a potential mechanism for VEGF-mediated vascular permeability in the eye. Similarly, in human non-ocular disease states such as ascites, VEGF has been characterized as a potent vascular permeability factor (VPF).

The normal human retina contains little or no VEGF; however, hypoxia causes upregulation of VEGF production. Vinores et al, using immunohistochemical staining for VEGF, demonstrated that increased VEGF staining was found in retinal neurons and retinal pigment epithelium in human eyes with diabetic retinopathy.

As the above discussion suggests, attenuation of the effects of VEGF provides a rationale for treatment of macular edema associated with diabetic retinopathy. Corticosteroids, a class of substances with anti-inflammatory properties, have been demonstrated to inhibit the expression of the VEGF gene. In a study by Nauck et al, the platelet-derived growth-factor (PDGF) induced expression of the VEGF gene in cultures of human aortic vascular smooth muscle cells was abolished by corticosteroids in a dose-dependent manner. A separate study by Nauck et al demonstrated that corticosteroids abolished the induction of VEGF by the pro-inflammatory mediators PDGF and platelet-activating factor (PAF) in a time and dose-dependent manner. This study was performed using primary cultures of human pulmonary fibroblasts and pulmonary vascular smooth muscle cells.

As discussed above, corticosteroids have been experimentally shown to down regulate VEGF production and possibly reduce breakdown of the blood-retinal barrier. Similarly, steroids have anti-angiogenic properties possibly due to attenuation of the effects of VEGF. Both of these steroid effects have been utilized. For example, triamcinolone acetonide is often used clinically as a periocular injection for the treatment of cystoid macular edema (CME) secondary to uveitis or as a result of intraocular surgery. In animal studies, intravitreal triamcinolone acetonide has been used in the prevention of proliferative vitreoretinopathy and retinal neovascularization. Intravitreal triamcinolone acetonide has been used clinically in the treatment of proliferative vitreoretinopathy and choroidal neovascularization.

ELIGIBILITY:
Subject Level Criteria Inclusion

To be eligible, the following inclusion criteria (1-4) must be met:

1. Age ≥18 years
2. Diagnosis of diabetes mellitus (type 1 or type 2)
3. At least one eye meets the study eye criteria
4. Able and willing to provide informed consent.

   Study Level Exclusion Criteria

   A patient is not eligible if any of the following exclusion criteria (5-13) are present:
5. History of chronic renal failure requiring dialysis or kidney transplant.
6. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control). Patients in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months should not be enrolled.
7. Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at the time of study entry.
8. Known allergy to any corticosteroid or any component of the delivery vehicle.
9. History of systemic (e.g., oral, IV, IM, epidural, bursal) corticosteroids within 4 months prior to randomization or topical, rectal, or inhaled corticosteroids in current use more than 2 times per week.
10. History of steroid-induced intraocular pressure elevation that required IOP-lowering treatment in either eye.
11. Warfarin (coumadin) currently being used.
12. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, patient can become eligible.
13. Patient is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the next 8 months.

    The patient must have at least one eye meeting all of the inclusion criteria (a-e) and none of the exclusion criteria (f-t) listed below:

    Study Eye Inclusion Criteria
    1. Best corrected electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity score of ≥69 letters (i.e., 20/40 or better).
    2. Definite retinal thickening due to diabetic macular edema based on clinical exam.
    3. Retinal thickness in the Optical Coherence Tomography (OCT) central subfield measuring 250 microns or more.
    4. Maximal laser has not already been given and investigator believes that either peribulbar steroids or laser may benefit the eye (note: subjects may be enrolled without having received prior macular laser).
    5. Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photographs and OCT.

       Study Eye Exclusion Criteria
    6. Macular edema is considered to be due to a cause other than diabetic macular edema.
    7. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, nonretinal condition).
    8. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc.).
    9. History of prior treatment with intravitreal, peribulbar, or retrobulbar corticosteroids for DME.
    10. History of focal/grid macular photocoagulation within 15 weeks (3.5 months) prior to randomization. Note: Patients are not required to have had prior macular photocoagulation to be enrolled.
    11. History of panretinal scatter photocoagulation (PRP) within 4 months prior to randomization or anticipated need for PRP in the 4 months following randomization.

    m. History of prior vitrectomy.

    n. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 6 months or anticipated within the next 6 months following randomization.

    o. History of YAG capsulotomy performed within 2 months prior to randomization.

    p. Intraocular pressure ≥25 mmHg.

    q. History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: angle-closure glaucoma is not an exclusion). A history of ocular hypertension is not an exclusion as long as (1) intraocular pressure is <25 mm Hg, (2) the patient is using no more than one topical glaucoma medication, (3) the most recent visual field, performed within the last 12 months, is normal (if abnormalities are present on the visual field they must be attributable to the patient's diabetic retinopathy), and (4) the optic disc does not appear glaucomatous. Note: if the intraocular pressure is 22 to <25 mm Hg, then the above criteria for ocular hypertension eligibility must be met.

    r. History of prior herpetic ocular infection.

    s. Exam evidence of ocular toxoplasmosis.

    t. Exam evidence of pseudoexfoliation.

    A patient may have two "study eyes" only if both are eligible at the time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-12; Primary Completion 2006-06 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chew, M.D., Study Chair — National Eye Institute (NEI)

REFERENCES:
- [Background] Chew EY, Glassman AR, Beck RW, Bressler NM, Fish GE, Ferris FL, Kinyoun JL; Diabetic Retinopathy Clinical Research Network. Ocular side effects associated with peribulbar injections of triamcinolone acetonide for diabetic macular edema. Retina. 2011 Feb;31(2):284-9. doi: 10.1097/IAE.0b013e3181f049a8. PMID 20948459
- [Result] Diabetic Retinopathy Clinical Research Network; Chew E, Strauber S, Beck R, Aiello LP, Antoszyk A, Bressler N, Browning D, Danis R, Fan J, Flaxel C, Friedman S, Glassman A, Kollman C, Lazarus H. Randomized trial of peribulbar triamcinolone acetonide with and without focal photocoagulation for mild diabetic macular edema: a pilot study. Ophthalmology. 2007 Jun;114(6):1190-6. doi: 10.1016/j.ophtha.2007.02.010. PMID 17544778
- [Derived] Gangaputra S, Almukhtar T, Glassman AR, Aiello LP, Bressler N, Bressler SB, Danis RP, Davis MD; Diabetic Retinopathy Clinical Research Network. Comparison of film and digital fundus photographs in eyes of individuals with diabetes mellitus. Invest Ophthalmol Vis Sci. 2011 Aug 3;52(9):6168-73. doi: 10.1167/iovs.11-7321. PMID 21571677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-two clinical sites across the United States recruited 129 eyes of 109 subjects between December 2004 and September 2005. 113 subjects were randomized, but 4 were not included in any of the analysis because they were ineligible.
Pre-assignment Details: Participants with two study eyes enrolled each eye in a different treatment group. Therefore, each treatment group/arm includes no more than one study eye for a given participant, and thus the numbers of eyes is equal to the number of participants in each arm.
Groups:
- Focal Laser Photocoagulation: Modified Early Treatment diabetic retinopathy Study technique (m-ETDRS, Laser burns-50 microns, gray intensity Multiple settings (all completed in single setting).
- Posterior Peribulbar Injection of 40 mg Triamcinolone: Posterior peribulbar injection of 40 mg triamcinolone (Kenalog)
- Anterior Peribulbar Injection of 20 mg Triamcinolone: Anterior peribulbar injection of 20 mg triamcinolone
- Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser: Posterior peribulbar injection of 40 mg triamcinolone followed by focal photocoagulation after one month
- Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser: Anterior peribulbar injection of 20 mg triamcinolone followed by focal photocoagulation after one month
Period: 4-Week Visit
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Started | 38 (Number of eyes) | 21 (Number of eyes) | 23 (Number of eyes) | 22 (Number of eyes) | 25 (Number of eyes)
Completed | 36 (Number of eyes) | 19 (Number of eyes;) | 22 (Number of eyes) | 20 (Number of eyes) | 24 (Number of eyes)
Not Completed | 2 | 2 | 1 | 2 | 1
Not completed — Missed visit | 2 | 2 | 0 | 2 | 1
Not completed — Dropped | 0 | 0 | 1 | 0 | 0
Period: 8-Week Visit
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Started | 38 (Number of eyes) | 21 (Number of eyes) | 22 (Number of eyes) | 22 (Number of eyes) | 25 (Number of eyes)
Completed | 38 (Number of eyes) | 20 (Number of eyes) | 22 (Number of eyes) | 21 (Number of eyes) | 24 (Number of eyes)
Not Completed | 0 | 1 | 0 | 1 | 1
Not completed — Missed visit | 0 | 1 | 0 | 0 | 1
Not completed — Dropped | 0 | 0 | 0 | 1 | 0
Period: 17-Week Visit
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Started | 38 (Number of eyes) | 21 (Number of eyes) | 23 (Number of eyes) | 22 (Number of eyes) | 25 (Number of eyes)
Completed | 38 (Number of eyes) | 21 (Number of eyes) | 22 (Number of eyes) | 21 (Number of eyes) | 24 (Number of eyes)
Not Completed | 0 | 0 | 1 | 1 | 1
Not completed — Missed visit | 0 | 0 | 1 | 1 | 1
Period: 34-Week Visit
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Started | 38 (Number of eyes) | 21 (Number of eyes) | 23 (Number of eyes) | 22 (Number of eyes) | 25 (Number of eyes that)
Completed | 38 (Number of eyes) | 20 (Number of eyes) | 22 (Number of eyes) | 19 (Number of eyes) | 22 (Number of eyes)
Not Completed | 0 | 1 | 1 | 3 | 3
Not completed — Dropped | 0 | 1 | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser | Total
Number analyzed (Participants) | 38 | 21 | 23 | 22 | 25 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11) | 58 (12) | 60 (8) | 64 (7) | 63 (13) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 5 | 4 | 8 | 47
  Male | 21 | 8 | 18 | 18 | 17 | 82
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31 | 16 | 21 | 19 | 19 | 106
  African-American | 3 | 3 | 0 | 3 | 4 | 13
  Hispanic or Latino | 1 | 1 | 2 | 0 | 1 | 5
  Asian | 3 | 1 | 0 | 0 | 0 | 4
  Other | 0 | 0 | 0 | 0 | 1 | 1
Cystoid Abnormality on Ocular Coherence Tomography (OCT) [Number; unit: eyes]
  Yes | 30 | 17 | 20 | 18 | 19 | 104
  No | 8 | 4 | 3 | 4 | 6 | 25
Diabetes Type [Number; unit: Participants]
  Type 1 | 3 | 3 | 3 | 0 | 1 | 10
  Type 2 | 35 | 18 | 20 | 22 | 24 | 119
Electronic Early Treatment Diabetic Retinopathy Study Visual Acuity [Number; unit: eyes] — Best corrected visual acuity letter score as measured by a certified tester using an electronic early treatment diabetic retinopathy study (e-ETDRS) method and approximate Snellen equivalent. Best value on the scale is 97, worst value 0.
  eyes
    >=79: 20/25 or better | 25 | 12 | 17 | 10 | 11 | 75
    78-69: 20/32-20/40 | 13 | 9 | 6 | 12 | 14 | 54
Received Prior Focal Photocoagulation [Number; unit: eyes]
  No | 21 | 7 | 8 | 10 | 11 | 57
  Yes | 17 | 14 | 15 | 12 | 14 | 72
Received Prior Scatter (Panretinal) Photocoagulation [Number; unit: eyes]
  No | 34 | 16 | 19 | 21 | 25 | 115
  Yes | 4 | 5 | 4 | 1 | 0 | 14
Subretinal Fluid on Ocular Coherence Tomography (OCT) [Number; unit: eyes] — Ocular Coherence Tomography (OCT) images were obtained at each visit following pupil dilation by a certified operator using the OCT3 machine (Carl Zeiss Meditec Inc., Dublin, CA). Scans were 6 mm length and included the 6 radial line pattern for quantitative measures and the cross hair pattern (6-12 to 9-3 o'clock) for qualitative assessment of retinal morphology.
  eyes
    Yes | 4 | 1 | 0 | 1 | 2 | 8
    No | 34 | 20 | 23 | 21 | 23 | 121
Central Subfield Thickness [Mean (Standard Deviation); unit: microns] — Measured by Ocular Coherence Tomography (OCT). OCT images were obtained at each visit following pupil dilation by a certified operator using the OCT3 machine (Carl Zeiss Meditec Inc., Dublin, CA). Scans were 6 mm length and included the 6 radial line pattern for quantitative measures and the cross hair pattern (6-12 to 9-3 o'clock) for qualitative assessment of retinal morphology.
  microns | 324 (70) | 321 (53) | 342 (79) | 319 (59) | 336 (58) | 328 (65)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — N=129 eyes
  years | 14 (10) | 14 (9) | 15 (7) | 16 (7) | 15 (9) | 15 (9)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage] | 7.9 (1.7) | 7.3 (1.6) | 8.1 (1.7) | 7.8 (1.3) | 7.5 (1.8) | 7.8 (1.6)
Intraocular Pressure (mm Hg) [Mean (Standard Deviation); unit: mm Hg] — N=129 eyes
  mm Hg | 16 (3) | 16 (4) | 16 (4) | 16 (3) | 17 (3) | 16 (3)
Mean visual acuity letter score [Mean (Standard Deviation); unit: letter score] — Baseline Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) Visual Acuity Letter Score: best value = 97; letter score worst value = 0
  letter score | 80 (5) | 79 (4) | 81 (5) | 79 (7) | 78 (6) | 79 (5)
Total Retinal Volume (mm^3) [Mean (Standard Deviation); unit: mm^3] | 8.2 (1.2) | 7.6 (0.9) | 8.1 (1.2) | 7.8 (0.6) | 7.9 (0.8) | 8.0 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Subfield Thickening From Baseline Through 34 Weeks
Description: Change in Central Subfield Thickening from Baseline measured on Optical Coherence Tomography (OCT). OCT images were obtained at each visit following pupil dilation by a certified operator using the OCT3 machine (Carl Zeiss Meditec Inc., Dublin, CA). Scans were 6 mm length and included the 6 radial line pattern for quantitative measures and the cross hair pattern (6-12 to 9-3 o'clock) for qualitative assessment of retinal morphology. Negative changes represent a decrease in retinal thickening.
Time Frame: 4, 8, 17, 34 weeks
Population: Last Observation Carried Forward was used. The correlation between eyes of patients who have two study eyes (one eye in the laser group and one eye in either of the Triamcinolone groups) was accounted for in the primary analysis. Primary analyses excluded patients who missed the visit.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Number analyzed (Participants) | 38 | 21 | 23 | 22 | 25
Number analyzed (Eyes) | 38 | 21 | 23 | 22 | 25
microns
  4 Weeks | -10 (53) | -47 (51) | -27 (36) | -16 (60) | -37 (66)
  8 Weeks | -27 (49) | -29 (62) | -38 (44) | -25 (55) | -44 (64)
  17 Weeks | -30 (60) | -24 (91) | -50 (49) | -52 (45) | -49 (79)
  34 Weeks | -54 (62) | -31 (113) | -45 (56) | -45 (70) | -68 (60)
Statistical Analysis 1: Comparison: Posterior Peribulbar Injection of 40 mg Triamcinolone vs Anterior Peribulbar Injection of 20 mg Triamcinolone vs Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser vs Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser; Comparison of change in central subfield thickening from baseline to 34 weeks in all five groups; Test type: Superiority or Other; p = 0.46, repeated measures least sq. regression — Adjusted for baseline central subfield thickness; Models adjusted for baseline values and for correlated data from subjects with two study eyes

2. Secondary Outcome: Persistence/Recurrence of Diabetic Macular Edema (DME) Either Retreated or Meeting Criteria for Retreatment at 17 Weeks
Description: Number of eyes that were retreated at 17 weeks. According to the protocol, primary criterion for retreatment was central subfield thickness >=250 microns or macular edema was still present according to the investigator's judgment.
Time Frame: 17 weeks
Population: The correlation between eyes of patients who have two study eyes (one eye in the laser group and one eye in either of the Triamcinolone groups) was accounted for in the primary analysis. Primary analyses excluded patients who missed the visit
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Number analyzed (Participants) | 38 | 21 | 22 | 21 | 24
Number analyzed (Eyes) | 38 | 21 | 22 | 21 | 24
eyes
  Eyes that were retreated | 22 | 15 | 14 | 9 | 9
  Eyes with ≥ 250 central subfield thickness | 26 | 14 | 16 | 11 | 13
Statistical Analysis 1: Comparison: Focal Laser Photocoagulation vs Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser vs Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser; Analysis combined posterior and anterior injection + laser groups to compare with laser only; Test type: Superiority or Other; p = 0.04, generalized estimating equations; Odds Ratio (OR) = 0.5, 95% CI [0.2 to 1.0]
Statistical Analysis 2: Comparison: Focal Laser Photocoagulation vs Posterior Peribulbar Injection of 40 mg Triamcinolone vs Anterior Peribulbar Injection of 20 mg Triamcinolone; Analysis combined posterior and anterior injection only groups to compare with laser only treatment group; Test type: Superiority or Other; p = 0.63, generalized estimating equations; Odds Ratio (OR) = 1.2, 95% CI [0.5 to 2.9]

3. Primary Outcome: Change in Visual Acuity Letter Score From Baseline Through 34 Weeks
Description: Change in visual acuity letter score as measured by a certified tester using an electronic visual acuity testing machine based on the electronic Early Treatment for Diabetic Retinopathy Study(E-ETDRS) technique. Letter score best value = 97 and worst value = 0; an increase in a letter score by 10 is considered clinically significant. Negative changes represent a worsening in visual acuity.
Time Frame: 4, 8, 17, and 34 weeks
Population: The primary analysis included all randomized eyes and followed the intent-to-treat analysis. The correlation between eyes of patients who have two study eyes (one eye in the laser group and one eye in either of the Triamcinolone groups) was accounted for in the primary analysis. Primary analyses excluded patients who missed the visit.
Measure: Mean (Standard Deviation); unit: letter score
Units Other Than Participants: Eyes
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Number analyzed (Participants) | 38 | 21 | 23 | 22 | 25
Number analyzed (Eyes) | 38 | 21 | 23 | 22 | 25
letter score
  4 Weeks | -1 (5) | 1 (4) | -1 (4) | -2 (6) | -1 (5)
  8 Weeks | -1 (5) | 0 (7) | -1 (6) | 0 (4) | 0 (6)
  17 Weeks | -2 (5) | -1 (6) | -2 (5) | -1 (7) | -1 (7)
  34 Weeks | -2 (12) | -4 (11) | -1 (5) | -3 (15) | -1 (7)
Statistical Analysis 1: Comparison: Focal Laser Photocoagulation vs Posterior Peribulbar Injection of 40 mg Triamcinolone vs Anterior Peribulbar Injection of 20 mg Triamcinolone vs Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser vs Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser; Comparison of the mean change in visual acuity letter score among the five groups at 34 weeks. Negative changes represent a worsening in visual acuity; Test type: Superiority or Other; p = 0.94, repeated measures least sq. regression; Adjusted for baseline values and for the correlated data from subjects with two study eyes

4. Primary Outcome: Mean Visual Acuity Letter Score at Each Follow-up Visit
Description: Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) mean visual acuity letter score: best value = 97; letter score worst value = 0
Time Frame: 4, 8, 17, and 34 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: letter score
Units Other Than Participants: Eyes
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Number analyzed (Participants) | 38 | 21 | 23 | 22 | 25
Number analyzed (Eyes) | 38 | 21 | 23 | 22 | 25
letter score
  4 Weeks | 79 (5) | 79 (5) | 80 (6) | 77 (7) | 77 (6)
  8 Weeks | 79 (5) | 79 (6) | 80 (7) | 80 (7) | 77 (6)
  17 Weeks | 78 (6) | 78 (5) | 79 (7) | 79 (7) | 77 (7)
  34 Weeks | 78 (12) | 76 (12) | 80 (8) | 77 (16) | 77 (7)

5. Secondary Outcome: Reduction of ≥ 50% in Retinal Thickening in the Central Subfield From Baseline Through 34 Weeks
Description: Number of eyes that had a reduction in central subfield retinal thickness by ≥ 50% at each follow-up. Change in Central Subfield Thickening from Baseline measured on Optical Coherence Tomography (OCT). OCT images were obtained at each visit following pupil dilation by a certified operator using the OCT3 machine (Carl Zeiss Meditec Inc., Dublin, CA). Scans were 6 mm length and included the 6 radial line pattern for quantitative measures and the cross hair pattern (6-12 to 9-3 o'clock) for qualitative assessment of retinal morphology.
Time Frame: 4, 8, 17, 34 weeks
Population: as for outcome 2
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Number analyzed (Participants) | 38 | 21 | 23 | 22 | 25
Number analyzed (Eyes) | 38 | 21 | 23 | 22 | 25
eyes
  4 Weeks | 5 | 8 | 2 | 4 | 8
  8 Weeks | 8 | 7 | 6 | 4 | 10
  17 Weeks | 11 | 6 | 8 | 7 | 13
  34 Weeks | 22 | 9 | 5 | 9 | 13

6. Secondary Outcome: Central Subfield Thickness <250 Microns From Baseline Through 34 Weeks
Description: Primary criterion for retreatment is central subfield thickness >=250 microns. Central subfield thickness of <250 microns indicates no need for retreatment. Change in Central Subfield Thickening from Baseline measured on Optical Coherence Tomography (OCT). OCT images were obtained at each visit following pupil dilation by a certified operator using the OCT3 machine (Carl Zeiss Meditec Inc., Dublin, CA). Scans were 6 mm length and included the 6 radial line pattern for quantitative measures and the cross hair pattern (6-12 to 9-3 o'clock) for qualitative assessment of retinal morphology.
Time Frame: 4, 8, 17, 34 weeks
Population: as for outcome 2
Measure: Number; unit: eyes
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Number analyzed (Participants) | 38 | 21 | 23 | 22 | 25
eyes
  4 Weeks | 5 | 5 | 3 | 2 | 8
  8 Weeks | 9 | 4 | 3 | 6 | 9
  17 Weeks | 11 | 7 | 6 | 10 | 11
  34 Weeks | 19 | 8 | 2 | 10 | 13

ADVERSE EVENTS:
Arm/Group | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Serious Adverse Events (participants affected / at risk) | 13 | 11 | 7 | 5 | 3
Other Adverse Events (participants affected / at risk) | 54 | 53 | 60 | 23 | 38
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Myocardial infarction (Cardiac disorders) | 0/38 | 1/21 | 0/23 | 3/22 | 0/25
Transient ischaemic attack (Cardiac disorders) | 0/38 | 0/21 | 0/23 | 2/22 | 0/25
Arteriosclerosis coronary artery (Cardiac disorders) | 0/38 | 0/21 | 1/23 | 0/22 | 0/25
Postoperative or localised infection (Infections and infestations) | 2/38 | 0/21 | 0/23 | 0/22 | 0/25
Cardiac operation (Cardiac disorders) | 0/38 | 0/21 | 0/23 | 0/22 | 1/25
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2/38 | 1/21 | 1/23 | 0/22 | 0/25
Heart failure (Cardiac disorders) | 1/38 | 0/21 | 0/23 | 0/22 | 0/25
Renal failure (Renal and urinary disorders) | 0/38 | 1/21 | 0/23 | 0/22 | 0/25
Multi-organ failure (General disorders) | 1/38 | 0/21 | 0/23 | 0/22 | 0/25
Fluid retention (General disorders) | 1/38 | 0/21 | 0/23 | 0/22 | 0/25
Skin ulcer or skin lesion (Skin and subcutaneous tissue disorders) | 1/38 | 0/21 | 2/23 | 0/22 | 0/25
Diabetic gastroparesis (Endocrine disorders) | 0/38 | 0/21 | 0/23 | 0/22 | 1/25
Dizziness (General disorders) | 0/38 | 0/21 | 1/23 | 0/22 | 0/25
Osteomyelities acute (Musculoskeletal and connective tissue disorders) | 1/38 | 0/21 | 0/23 | 0/22 | 0/25
Oxygen saturation decreased (General disorders) | 1/38 | 0/21 | 0/23 | 0/22 | 0/25
Anaemia (Blood and lymphatic system disorders) | 1/38 | 1/21 | 0/23 | 0/22 | 0/25
Artery occlusion (Cardiac disorders) | 0/38 | 2/21 | 1/23 | 0/22 | 0/25
Chest discomfort (Cardiac disorders) | 1/38 | 0/21 | 0/23 | 0/22 | 0/25
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0/38 | 1/21 | 0/23 | 0/22 | 0/25
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0/38 | 2/21 | 0/23 | 0/22 | 0/25
Amputation (Surgical and medical procedures) | 0/38 | 0/21 | 1/23 | 0/22 | 0/25
Pulmonary embolism (Cardiac disorders) | 0/38 | 1/21 | 0/23 | 0/22 | 0/25
Cerebrovascular accident (Cardiac disorders) | 1/38 | 0/21 | 0/23 | 0/22 | 1/25
Gastric ulcer (Gastrointestinal disorders) | 0/38 | 1/21 | 0/23 | 0/22 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Focal Laser Photocoagulation | Posterior Peribulbar Injection of 40 mg Triamcinolone | Anterior Peribulbar Injection of 20 mg Triamcinolone | Posterior Peribulbar Injection of 40 mg Triamcinolone + Laser | Anterior Peribulbar Injection of 20 mg Triamcinolone + Laser
Ptosis (Eye disorders) | 0/38 (0) | 4/21 | 3/23 | 1/22 | 1/25
Elevated intraocular pressure/glaucoma (increase by 10mm Hg or more at any visit) (Eye disorders) | 2/38 | 3/21 | 10/23 | 5/22 | 13/25
HbA1c (increase by 0.5% or more from baseline) (Endocrine disorders) | 11/38 | 5/21 | 8/23 | 5/22 | 6/25
Cataract (Eye disorders) | 3/38 | 2/21 | 4/23 | 1/22 | 5/25
Cataract cortical (Eye disorders) | 1/38 | 1/21 | 2/23 | 2/22 | 0/25
Cataract subcapsular (Eye disorders) | 2/38 | 1/21 | 3/23 | 2/22 | 2/25
Conjunctival haemorrhage (Eye disorders) | 0/38 | 5/21 | 9/23 | 0/22 | 1/25
Diabetic retinopathy (Endocrine disorders) | 3/38 | 2/21 | 0/23 | 0/22 | 1/25
Eye pain (Eye disorders) | 0/38 | 3/21 | 1/23 | 0/22 | 1/25
Lacrimation increased (Eye disorders) | 0/38 | 2/21 | 0/23 | 0/22 | 0/25
Vision blurred (Eye disorders) | 2/38 | 3/21 | 1/23 | 1/22 | 1/25
Visual acuity reduced (Eye disorders) | 0/38 | 1/21 | 1/23 | 2/22 | 3/25
Visual disturbance (Eye disorders) | 3/38 | 5/21 | 0/23 | 4/22 | 1/25
Vitreous floaters (Eye disorders) | 2/38 | 0/21 | 0/23 | 0/22 | 1/25
Vitreous haemorrhage (Eye disorders) | 7/38 | 0/21 | 0/23 | 0/22 | 0/25
Subconjunctival haemorrhage (Eye disorders) | 0/38 | 0/21 | 3/23 | 0/22 | 1/25
Anaemia (Blood and lymphatic system disorders) | 2/38 | 2/21 | 0/23 | 0/22 | 0/25
Arteriosclerosis coronary artery (Cardiac disorders) | 0/38 | 0/21 | 2/23 | 0/22 | 0/25
Cough (Respiratory, thoracic and mediastinal disorders) | 1/38 | 0/21 | 3/23 | 0/22 | 0/25
Diarrhoea (Gastrointestinal disorders) | 0/38 | 2/21 | 1/23 | 0/22 | 0/25
Gastric ulcer (Gastrointestinal disorders) | 0/38 | 3/21 | 0/23 | 0/22 | 0/25
Hypercholesterolaemia (Cardiac disorders) | 2/38 | 1/21 | 1/23 | 0/22 | 0/25
Hyperlipidaemia (Cardiac disorders) | 2/38 | 1/21 | 1/23 | 0/22 | 0/25
Hypertension (Cardiac disorders) | 2/38 | 1/21 | 2/23 | 0/22 | 1/25
Limb injury (Musculoskeletal and connective tissue disorders) | 0/38 | 2/21 | 0/23 | 0/22 | 0/25
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2/38 | 0/21 | 0/23 | 0/22 | 0/25
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0/38 | 2/21 | 0/23 | 0/22 | 0/25
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2/38 | 1/21 | 1/23 | 0/22 | 0/25
Skin ulcer (Skin and subcutaneous tissue disorders) | 2/38 | 1/21 | 1/23 | 0/22 | 0/25
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1/38 | 0/21 | 2/23 | 0/22 | 0/25
Urinary tract infection (Renal and urinary disorders) | 2/38 | 0/21 | 1/23 | 0/22 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No